CLINICAL TRIAL: NCT02187068
Title: Dexmedetomidine Pharmacokinetics in the Obese
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 11-142
Record Dates: First submitted 2014-06-25; First posted 2014-07-10 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Obesity
Keywords: Anaesthetics iv; Dexmedetomidine; Pharmacokinetic
MeSH Terms: conditions — Obesity | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dexmedetomidine obese 1 (Experimental): 10 obese patients scheduled for elective laparoscopic surgery were given dexmedetomidine dexmedetomidine 0.5 μg.kg-1 iv over 10 minutes and then dexmedetomidine 0.25 mcg.kg-1.h-1 for approximate 2 h (range 58-320 min). Blood samples were taken at 2, 5, 10, 15, 20, 30, 45, 60, 90, 120 min after beginning dexmedetomidine administration, and at 0, 2, 5, 10, 20, 30, 60, 90, 120, 240 and 360 min after stopping infusion.
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine obese 2 (Experimental): 10 obese patients scheduled for elective laparoscopic surgery were given dexmedetomidine dexmedetomidine 0.5 μg.kg-1 iv over 10 minutes and then dexmedetomidine 0.5 mcg.kg-1.h-1 for approximate 2 h (range 58-320 min). Blood samples were taken at 2, 5, 10, 15, 20, 30, 45, 60, 90, 120 min after beginning dexmedetomidine administration, and at 0, 2, 5, 10, 20, 30, 60, 90, 120, 240 and 360 min after stopping infusion.
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine non-obese 1 (Experimental): 10 non-obese patients scheduled for elective laparoscopic surgery were given dexmedetomidine dexmedetomidine 0.5 μg.kg-1 iv over 10 minutes and then dexmedetomidine 0.25 mcg.kg-1.h-1 for approximate 2 h (range 58-320 min). Blood samples were taken at 2, 5, 10, 15, 20, 30, 45, 60, 90, 120 min after beginning dexmedetomidine administration, and at 0, 2, 5, 10, 20, 30, 60, 90, 120, 240 and 360 min after stopping infusion.
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine non obese 2 (Experimental): 10 non-obese patients scheduled for elective laparoscopic surgery were given dexmedetomidine dexmedetomidine 0.5 μg.kg-1 iv over 10 minutes and then dexmedetomidine 0.5 mcg.kg-1.h-1 for approximate 2 h (range 58-320 min). Blood samples were taken at 2, 5, 10, 15, 20, 30, 45, 60, 90, 120 min after beginning dexmedetomidine administration, and at 0, 2, 5, 10, 20, 30, 60, 90, 120, 240 and 360 min after stopping infusion.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine administered intravenously
  Other Names: Other names:; Precedex

SUMMARY:
The aim of this study is to characterize, using two different modeling approaches, one based on purely statistic concept and one using a more mechanistic analysis, the influence of body weight and composition on the pharmacokinetic of dexmedetomidine.

DETAILED DESCRIPTION:
Twenty obese patients and 20 non-obese patients scheduled for elective laparoscopic surgery will give dexmedetomidine 0.5 μg.kg-1 over 10 minutes and then randomized to either dexmedetomidine 0.25 mcg.kg-1.h-1 or dexmedetomidine 0.5 mcg.kg-1.h-1 for approximate 2 h (range 58-320 min). Blood samples will be taken at 2, 5, 10, 15, 20, 30, 45, 60, 90, 120 min after beginning dexmedetomidine administration, and at 0, 2, 5, 10, 20, 30, 60, 90, 120, 240 and 360 min after stopping infusion. Population pharmacokinetic modeling will be performed using nonlinear mixed-effects model.

ELIGIBILITY:
Inclusion Criteria:

* American Society Anesthesiologist classification I-III patients
* between 18 and 60 years of age
* scheduled for elective laparoscopic surgery
* obese patients with a BMI >35 kg m-2 (20 patients)
* non-obese patients (BMI 18.5-25 kg m-2)(20 patients)

Exclusion Criteria:

* known allergy to study drugs
* uncontrolled hypertension
* heart block greater than first degree
* those who had taken any drug acting in the central nervous system 24 h before surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
dexmedetomidine serum concentration | During the intraoperative period and 360 min after stopping dexmedetomidine infusion
  A two compartment distribution model with first order elimination was used to describe dexmedetomidine serum concentration. Population parameter estimates were obtained using non-linear mixed effects models

CONTACTS AND LOCATIONS:
Overall Officials: Luis I Cortínez, MD, Principal Investigator — Departamento de Anestesiología, Hospital Clínico Pontificia Universidad Católica de Chile
Locations (1):
- Hospital Clinico Pontificia Universidad Catolica, Santiago, Santiago Metropolitan, Chile